CLINICAL TRIAL: NCT07091851
Title: A Hybrid Type 1 Randomized Trial for Improved Post-Stroke Hypertension: This Study Aims to Examine the Impact of Group Medical Visits and Home Blood Pressure Monitoring Versus Home Blood Pressure Monitoring Alone on the the Impact of Hypertension in Those With Recent Stroke.
Brief Title: BRIDGE: Blood Pressure Reduction and Intervention Delivery Via Group Engagement
Acronym: BRIDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Nirupama Yechoor, MD, MSC, Instructor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025P001538
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hypertension; Home Blood Pressure Monitoring; Implementation Research
Keywords: stroke; post-stroke hypertension; implementation science
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Active Comparator): Home blood pressure monitoring alone
  Interventions: Behavioral: Group medical visits and home blood pressure monitoring

INTERVENTIONS:
Behavioral: Group medical visits and home blood pressure monitoring — This arm will receive instructions for home blood pressure monitoring but also be enrolled in group medical visits.

SUMMARY:
The investigators want to improve care for people who have had a stroke. High blood pressure is the leading cause for having a second stroke and can lead to poor brain health. The goal of this study is to compare two new ways of lowering blood pressure. The first way is to help people check their blood pressure at home. The second way is to bring people together and learn about blood pressure in a group setting. The study team thinks that using both methods together will make it easier to lower blood pressure after a stroke. The study team needs this study to test these two methods together in people who have had a stroke. The investigators believe this is an important study because having high blood pressure makes having another stroke very likely. Therefore, the investigators want to lower blood pressure in people with strokes to keep their brains as healthy as possible and to help with stroke recovery.

DETAILED DESCRIPTION:
Lowering blood pressure is a clear and effective target for improved secondary stroke prevention. Two evidenced-based interventions have shown clinical effectiveness in non-stroke populations to improve hypertension. Frist, home blood pressure monitoring (HBPM) has been shown to be accurate, pragmatic, effective, and incorporated into AHA guidelines. The second evidence-based intervention is the virtual group visit (VGV) model. VGVs are shared medical appointments conducted over virtual conference rooms that aim to provide pragmatic, patient-centered, cost-effective care for chronic disease management by leveraging patients' shared lived experiences to create a supportive community. The study team's prior studies show that VGVs that incorporate HBPM are feasible and effective in a prospective cohort of primary care patients. The investigators have generated preliminary data also suggest that stroke survivors find serial virtual focus groups feasible and useful. However, no studies to date have tested VGVs that incorporate HBPM in a stroke survivor population. The long-term goal of this proposal is to use implementation science to investigate alternative models of care to promote neuro-recovery and improve secondary stroke prevention. The overall research objective of this proposal is to first adapt existing evidence-based interventions using the CFIR framework, then conduct a Hybrid Type 1 randomized control trial to test effectiveness of a VGV-HBPM intervention compared to HBPM-alone in stroke survivors, and finally to measure the implementation outcomes of adoption and acceptability using the RE-AIM framework. The central hypothesis is that a VGV-HBPM intervention will result in superior BP control at 3-months compared to HBPM-alone in stroke survivors and will have high adoption and acceptability.

The rationale for this proposed research is that two evidence-based interventions show promise to help lower blood pressure and could be adapted for a very high-risk patient population. Guided by proven implementation science frameworks, three aims will be investigated: 1) adapt a VGV-HBPM model for stroke survivors and caregivers; 2) conduct a pilot randomized control trial to test the effectiveness of VGV-HBPM compared to HBPM-alone in stroke survivors; 3) measure the adoption and acceptability of our intervention. Successful completion of this proposal will lead to a refined, implementation-ready intervention and inform a fully powered efficacy trial for future proposals.

ELIGIBILITY:
Inclusion Criteria:

* Incident, mild to moderate, ischemic or hemorrhagic stroke (NIHSS≤15, ICH score≤3)
* history or new diagnosis of hypertension
* ability to read and speak English
* internet access
* established primary care physician at MGH

Exclusion Criteria:

* severe stroke (NIHSS>15, ICH score>3)
* discharge location to inpatient rehabilitation or skilled nursing facility
* dementia
* subjects with moderate to severe aphasia without a caregiver to consent on their behalf

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | three months
  mean systolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No